CLINICAL TRIAL: NCT01130519
Title: A Phase II Study of Bevacizumab and Erlotinib in Subjects With Advanced Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC) or Sporadic Papillary Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ramaprasad Srinivasan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100114; 10-C-0114
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: HLRCC; Sporadic Papillary Renal Cell Cancer
Keywords: Immunotherapy; Biomarker; Kidney Cancer; Renal Cell Cancer; Hereditary Leiomyomatosis and Renal Cell Cancer; HLRCC
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Hereditary leiomyomatosis and renal cell cancer | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 - Bevacizumab and Erlotinib (Experimental): All patients will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO)
  Interventions: Drug: Bevacizumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Bevacizumab — Commercially available. Administered by intravenous infusion.
  Other Names: Avastin
Drug: Erlotinib — Commercially available. Administered orally.
  Other Names: Tarceva

SUMMARY:
Background:

* At the present time, there are no drugs that have been proven to work in patients with papillary kidney cancer that has spread (metastasized) beyond the kidneys. Researchers are interested in determining whether the combination of the drugs bevacizumab and erlotinib can be used to treat metastatic papillary kidney cancer.
* Hereditary Leiomyomatosis and Renal Cell Carcinoma (HLRCC) is an inherited type of papillary kidney cancer (it runs in families). Papillary kidney cancer can also occur sporadically, or without a family connection. More research is needed to determine whether treatments for papillary kidney cancer, such as bevacizumab and erlotinib, work in inherited or sporadic types of kidney cancer, and if so, whether there are any differences.

Objectives:

-To determine the effectiveness of the combination of bevacizumab and erlotinib as a treatment for patients with (1) metastatic HLRCC kidney cancer and (2) metastatic kidney cancer not associated with HLRCC (or sporadic papillary RCC).

Eligibility:

* Individuals 18 years of age or older who have been diagnosed with papillary kidney cancer that has spread beyond the kidneys.
* Participants may have either HLRCC or sporadic papillary kidney cancer.

Design:

* Participants will be screened with a full medical history, physical examination, blood and urine tests, and computed tomography (CT) and other scans to evaluate tumor size and treatment options.
* Participants will receive 28-day treatment cycles of bevacizumab (given intravenously every 2 weeks) and erlotinib (a tablet taken by mouth daily).
* Every cycle, participants will return for regular blood and urine tests. Every other cycle, participants will have imaging scans to assess tumor size and response to treatment. Female participants who have uterine fibroid tumors related to their kidney cancer may have additional scans to assess tumor size and response to treatment.
* Participants will continue to receive treatment on the study until their tumors grow or spread to new areas (disease progression), intolerable side effects develop, a better treatment option becomes available, the study closes, it is unsafe to continue treatment, or the participant decides not to remain in the study.

DETAILED DESCRIPTION:
Background

* Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC) is a familial cancer syndrome characterized by a propensity for developing renal cancer, and uterine and cutaneous leiomyomas. The kidney cancer associated with HLRCC is clinically aggressive and is characterized by unique histopathologic features that are sometimes described as type 2 papillary RCC.
* Germline mutations in the fumarate hydratase (FH) gene are the genetic hallmark of HLRCC. Mutational inactivation of FH has been shown to result in Von Hippel-Lindau (VHL)-independent upregulation of hypoxia inducible factor (HIF) and its downstream transcriptional targets.
* The recognition that HIF upregulation may play an important role in the formation and propagation of renal cancer associated with HLRCC suggests that interventions directed against components of this pathway, such as vascular endothelial growth factor (VEGF) and transforming growth factor-alpha/epidermal growth factor receptor (EGFR), may be of benefit in this patient population.
* We propose to test the hypothesis that dual VEGF/EGFR blockade with bevacizumab/erlotinib is likely to be clinically active in patients with HLRCC associated RCC as well as those with sporadic papillary sporadic RCC.

Objective

Primary Objective

-To determine the overall response rate (Response Evaluation Criteria in Solid Tumors (RECIST) in patients with 1) metastatic RCC associated with HLRCC and 2) metastatic sporadic/non-HLRCC papillary renal cancer treated with a combination of bevacizumab and erlotinib

Eligibility

* Diagnosis of advanced RCC associated with HLRCC (cohorts 1 and 3) or sporadic/non-HLRCC papillary RCC (cohorts 2 and 4)
* Eastern Cooperative Oncology Group (ECOG) PS 0-2
* Measurable disease, consistent with RECIST 1.1
* No history of major bleeding, recent or active myocardial ischemia, gastrointestinal (GI) perforation, cerebrovascular accidents or other significant intercurrent illness
* No coagulopathy or bleeding diathesis
* No recent surgery (< 4 weeks or inadequately healed surgical scars)
* Adequate organ function
* Adequate liver function (total bilirubin <= 1.5 mg/dL or < 3 x upper limit of normal (ULN) in subjects with Gilbert's disease, and aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transferase (SGPT) 2.5 x ULN
* Adequate renal function (creatinine <= 2.0 x ULN or creatinine clearance > 30 mL/min
* Neutrophils >1500/microL and platelets >100,000
* No brain metastases
* No more than 2 prior regimens containing a VEGF-pathway inhibitor; no prior therapy with bevacizumab
* Ability to understand and sign informed consent

Design

* Patients will receive a fixed starting dose of bevacizumab (10mg/kg intravenous (IV) every 2 weeks) and erlotinib (150mg/day by mouth (po). Dose reductions and drug interruptions for unacceptable toxicity will be allowed.
* Patients will be evaluated for response every 8 weeks using RECIST criteria
* The study is based on an open label Simon two-stage minmax design in two cohorts, 1) cohort 1- patients with HLRCC, and 2) cohort 2- patients with sporadic papillary RCC. In each cohort, 13 patients will be accrued in the first stage and will accrue a maximum of 20 patients. Accrual into and analysis of the two cohorts will be independent.
* Following completion of accrual to cohorts 1 and 2, the study was expanded to include two additional cohorts- Cohort 3 (HLRCC patients and Cohort 4 (patients with sporadic/non HLRCC papillary RCC) to better estimate the overall response rate and to perform additional exploratory biomarker analyses. Up to 20 additional evaluable patients will be included in each of these cohorts.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must meet all the following criteria to be eligible for study enrolment:

* Diagnosis of advanced renal cell cancer (RCC) associated with hereditary leiomyomatosis and renal cell cancer (HLRCC) (cohorts 1 & 3) or sporadic/non-HLRCC papillary RCC (cohort 2 & 4)
* Measurable disease outlined in Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* No more than two prior regimens targeting the vascular endothelial growth factor (VEGF) pathway; no prior bevacizumab therapy
* Age greater than or equal to 18 years.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients must have normal organ and marrow function as defined below: white blood cell (WBC) count greater than or equal to 3,000/microL, absolute neutrophil count greater than or equal to 1,500/microL, platelet count greater than or equal to 100,000/microL, serum creatinine greater than or equal to 2 times the upper limit of reference range or creatinine clearance greater than or equal to 30 ml/min, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times the upper limit of reference range, total bilirubin less than 1.5 times the upper limit of reference range ( less than 3 x upper limit of reference range in patients with Gilbert's disease), alkaline phosphatase less than or equal to 2.5 times the upper limit of reference range (or less than or equal to 5 times the upper limit of reference range if considered to be related to liver or bone metastases by the principal investigator (PI)
* Recovery from acute toxicity of prior treatment for RCC (to less than or equal to grade 1 the active version of Common Terminology Criteria for Adverse Events (CTCAE) or to a level permitted under other sections of Inclusion/ Exclusion criteria).
* At least 4 weeks from completion of major surgery and a healed surgical incision
* Negative pregnancy test (within 7 days of enrolment) in women of childbearing potential
* No myocardial infarction, gastrointestinal (GI) perforation/fistula, intra-abdominal abscess, cerebrovascular accidents within six months prior to study entry
* No coagulopathy or bleeding diathesis
* Ability to understand and the willingness to sign a written informed consent document.
* Archival tissue block or unstained tumor tissue available for correlative studies

EXCLUSION CRITERIA:

* Prior invasive malignancy of other histology, with the exception of adequately treated basal or squamous cell carcinoma of the skin, or any other malignancy for which the patient does not currently require treatment and/or has no evidence of disease for greater than or equal to 2 years.
* Patients with known brain metastases unless treated with an appropriate modality with no evidence of progression/recurrence for greater than 3 months
* Hypertension not controlled by medical therapy (resting systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg on at least two occasions over a 24 hour period despite optimal medical management).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure (New York Heart Association grade III or greater), unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Serious, non-healing wound or ulcer; bone fracture within 3 months prior to study entry
* Patient known to be human immunodeficiency virus (HIV)-positive and requiring antiretroviral therapy (due to the risk of potential drug interactions)
* Concomitant therapy with potent inhibitors of Cytochrome P450 3A4 (CYP450 3A4) (e.g., ketoconazole, verapamil etc.) or with potent CYP450 1A2 inhibitors (fluoroquinolone antibiotics including ciprofloxacin, levofloxacin, and norfloxacin; ticlodipine, cimetidine, amiodarone, etc. see Appendix C)
* Pregnant women are excluded from this study because bevacizumab and erlotinib are anti-cancer agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on this study
* All men and women of childbearing potential must be willing to use effective contraception as determined by the principal investigator (including but not limited to abstinence, hormonal contraceptives (birth control pills, injections, or implants), intrauterine device (IUD), tubal ligation, vasectomy) from the time of enrolment to at least six months following the last dose of drug
* Any known hypersensitivity to bevacizumab, erlotinib or other excipients of these drugs
* Documented baseline proteinuria greater than 1000mg/day on 24-hour urine collection. Only patients with 1+ or greater proteinuria on urinalysis (UA) and a spot urine protein: creatinine ratio of greater than 0.5 will undergo a 24-hour urine collection for quantitation of proteinuria.
* Left ventricular ejection fraction less than 40% as measured on transthoracic echocardiogram.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-05-06 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Wei MH, Toure O, Glenn GM, Pithukpakorn M, Neckers L, Stolle C, Choyke P, Grubb R, Middelton L, Turner ML, Walther MM, Merino MJ, Zbar B, Linehan WM, Toro JR. Novel mutations in FH and expansion of the spectrum of phenotypes expressed in families with hereditary leiomyomatosis and renal cell cancer. J Med Genet. 2006 Jan;43(1):18-27. doi: 10.1136/jmg.2005.033506. Epub 2005 Jun 3. PMID 15937070
- [Background] Lehtonen HJ, Kiuru M, Ylisaukko-Oja SK, Salovaara R, Herva R, Koivisto PA, Vierimaa O, Aittomaki K, Pukkala E, Launonen V, Aaltonen LA. Increased risk of cancer in patients with fumarate hydratase germline mutation. J Med Genet. 2006 Jun;43(6):523-6. doi: 10.1136/jmg.2005.036400. Epub 2005 Sep 9. PMID 16155190
- [Background] Merino MJ, Torres-Cabala C, Pinto P, Linehan WM. The morphologic spectrum of kidney tumors in hereditary leiomyomatosis and renal cell carcinoma (HLRCC) syndrome. Am J Surg Pathol. 2007 Oct;31(10):1578-85. doi: 10.1097/PAS.0b013e31804375b8. PMID 17895761
- [Derived] Srinivasan R, Gurram S, Singer EA, Sidana A, Al Harthy M, Ball MW, Friend JC, Mac L, Purcell E, Vocke CD, Ricketts CJ, Kong HH, Cowen EW, Malayeri AA, Shih JH, Merino MJ, Linehan WM. Bevacizumab and Erlotinib in Hereditary and Sporadic Papillary Kidney Cancer. N Engl J Med. 2025 Jun 19;392(23):2346-2356. doi: 10.1056/NEJMoa2200900. PMID 40532152
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0114.html

RESULTS

PARTICIPANT FLOW:
Groups:
- COHORT 1-Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis and Renal Cell Cancer; COHORT 3 - Hereditary Leiomyomatosis and Renal Cell Cancer Associated Kidney Cancer: All participants will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO).
  Participants with metastatic Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC), diagnosed by either germline mutation of the fumarate hydratase (FH) gene, or based upon evidence of the clinical syndrome of HLRCC (characteristic renal cancer histology, cutaneous leiomyomas, uterine fibroids, and a family history).
- COHORT 2 - Sporadic Papillary Renal Cell Cancer; COHORT 4-Sporadic/NonHereditary Leiomyomatosis and Renal Cell Cancer Papillary Kidney Cancer: All participants will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO).
  Participants with sporadic papillary renal cancer.
Period: Overall Study
Arm/Group | COHORT 1-Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis and Renal Cell Cancer | COHORT 2 - Sporadic Papillary Renal Cell Cancer | COHORT 3 - Hereditary Leiomyomatosis and Renal Cell Cancer Associated Kidney Cancer | COHORT 4-Sporadic/NonHereditary Leiomyomatosis and Renal Cell Cancer Papillary Kidney Cancer
Started | 20 | 21 | 23 | 19
Completed | 20 | 21 | 23 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COHORT 1-Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis and Renal Cell Cancer | COHORT 2 - Sporadic Papillary Renal Cell Cancer | COHORT 3 - Hereditary Leiomyomatosis and Renal Cell Cancer Associated Kidney Cancer | COHORT 4-Sporadic/NonHereditary Leiomyomatosis and Renal Cell Cancer Papillary Kidney Cancer | Total
Number analyzed (Participants) | 20 | 21 | 23 | 19 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 22 | 16 | 74
  >=65 years | 0 | 5 | 1 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.43 (12.15) | 56.99 (9.61) | 44.53 (12.98) | 52.37 (13.98) | 49.21 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 3 | 8 | 27
  Male | 10 | 15 | 20 | 11 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 19 | 20 | 22 | 19 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 1 | 4
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 1 | 3 | 8
  White | 15 | 21 | 20 | 15 | 71
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 23 | 19 | 83

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Participants whose tumors regressed (Complete Response (CR) plus Partial Response (PR)) after therapy as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the longest diameters of target lesions. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Data shown with 95% confidence intervals.
Time Frame: Every 8 weeks during the first 32 weeks and every 12 weeks thereafter, a median of 64.3 months
Population: As pre-specified by the protocol for reporting purposes, our expansion cohorts were combined with the original cohorts (i.e., cohort 1, cohort 2, cohort 3, and cohort 4). Therefore, we reported on two groups: all Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC) participants (Cohorts 1 & 3) and all sporadic participants (Cohort 2 & 4).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer: COHORT 1 - Advanced Renal Cell Cancer Associated with Hereditary Leiomyomatosis and Renal Cell Cancer
  All participants will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO).
  Participants with metastatic Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC), diagnosed by either germline mutation of the fumarate hydratase (FH) gene, or based upon evidence of the clinical syndrome of HLRCC (characteristic renal cancer histology, cutaneous leiomyomas, uterine fibroids, and a family history).
  COHORT 3 - Hereditary Leiomyomatosis and Renal Cell Cancer Associated Kidney Cancer
  All participants will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO).
  Participants with metastatic Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC), diagnosed by either germline mutation of the fumarate hydratase (FH) gene, or based upon evidence of the clinical syndrome of HLRCC (characteristic renal cancer histology, cutaneous leiomyomas, uterine fibroids, and a family history).
- COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer: COHORT 2 - Sporadic Papillary Renal Cell Cancer
  All participants will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO).
  Participants with sporadic papillary renal cancer.
  COHORT 4 - Sporadic/NonHereditary Leiomyomatosis and Renal Cell Cancer Papillary Kidney Cancer
  All participants will be receiving fixed starting dose of bevacizumab (10 mg/kg intravenous (IV) every 2 weeks) and erlotinib (150 mg/day by mouth (PO).
  Participants with sporadic papillary renal cancer.
Arm/Group | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer
Number analyzed (Participants) | 43 | 40
Percentage of participants | 72 [57 to 83] | 35 [22 to 51]

2. Secondary Outcome: Progression-free Survival
Description: Median amount of time subject survives without disease progression after treatment. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Amount of time subject survives without disease progression after treatment; a median of 15 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer
Number analyzed (Participants) | 43 | 40
Months | 21.1 [15.6 to 26.6] | 8.9 [5.5 to 18.3]

3. Secondary Outcome: Duration of Response
Description: Duration of overall response is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started), measured by the Response Evaluation Criteria in Solid Tumors (RECIST). CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented; a median of 19 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer
Number analyzed (Participants) | 43 | 40
Months | 19.3 [12.9 to 35.9] | 18.4 [13.8 to 49.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the duration of time from the date of study enrolment until time of death estimated using a Kaplan Meier analysis. Participants without a death event will be censored at the date survival assessment was last evaluated (e.g., clinic visit, phone call).
Time Frame: Time from the date of study enrolment until time of death; a median of 29.3 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer
Number analyzed (Participants) | 43 | 40
Months | 44.6 [32.7 to NA] — Because the upper limit of the Kaplan-Meier curve for OS in the HLRCC cohorts hasn't reached 50%, there is no estimate for the upper confidence limit on the median. As such, we report the upper bound of the 95% CI as not estimable. | 18.2 [12.6 to 29.3]

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 133 months and 13 days; and 119 months and 2 days for the first and second group respectively.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer
Number analyzed (Participants) | 43 | 40
Participants | 43 | 40

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 133 months and 13 days; and 119 months and 2 days for the first and second group respectively.
Description: As pre-specified by the protocol for safety/adverse events reporting purposes, expansion cohorts were combined with original cohorts (cohort 1-4). Thus, we reported on 2 groups: all Hereditary Leiomyomatosis and Renal Cell Cancer participants (Cohorts 1&3) and all sporadic participants (Cohort 2&4). Participants whose survival was obtained from other publicly available data sources/other National Institutes of Health protocols in which participants are co-enrolled are included in mortality.
Arm/Group | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer
All-Cause Mortality (participants affected / at risk) | 28/43 | 36/40
Serious Adverse Events (participants affected / at risk) | 9/43 | 9/40
Other Adverse Events (participants affected / at risk) | 43/43 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer (N=43) | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Migraine headache (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1&3 Advanced Renal Cell Cancer Associated With Hereditary Leiomyomatosis & Renal Cell Cancer (N=43) | COHORT 2 and 4 - Sporadic Papillary Renal Cell Cancer (N=40)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 15 (24) | 6 (10)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Akathisia (Nervous system disorders) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 16 (46) | 18 (39)
Alkaline phosphatase increased (Investigations) | 7 (20) | 17 (33)
Allergic reaction (Immune system disorders) | 1 (2) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (18) | 12 (12)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 14 (45) | 9 (13)
Anorexia (Metabolism and nutrition disorders) | 10 (17) | 14 (19)
Anxiety (Psychiatric disorders) | 4 (6) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 22 (73) | 19 (56)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 8 (16)
Bladder infection (Infections and infestations) | 2 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 4 (7) | 3 (3)
Blood and lymphatic system disorders - Other, Iron deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 11 (34) | 14 (59)
Blurred vision (Eye disorders) | 3 (4) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CPK increased (Investigations) | 23 (117) | 10 (29)
Cardiac disorders - Other, Postural Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (4) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (11) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (30) | 20 (26)
Creatinine increased (Investigations) | 31 (171) | 17 (79)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
Dental caries (Gastrointestinal disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 11 (14) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 40 (112) | 34 (77)
Dizziness (Nervous system disorders) | 9 (15) | 7 (11)
Dry eye (Eye disorders) | 5 (6) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (32) | 23 (25)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 15 (19) | 15 (18)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 4 (4)
Ear and labyrinth disorders - Other, Clogged ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 6 (9) | 3 (4)
Edema trunk (General disorders) | 4 (5) | 2 (2)
Endocrine disorders - Other, Drenching night sweats (Endocrine disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other, Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 (43) | 12 (14)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Blepharitis (Eye disorders) | 3 (4) | 1 (1)
Eye disorders - Other, Eye Pressure R eye (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, Eyelash growth (Eye disorders) | 3 (3) | 0 (0)
Eye disorders - Other, Eyelid spasm (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, L eye scleral hematoma (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Stye on L eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Styes in bilat upper eyelid (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Fatigue (General disorders) | 23 (60) | 25 (39)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 2 (2) | 7 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (6)
Flatulence (Gastrointestinal disorders) | 4 (4) | 2 (2)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 9 (13) | 4 (4)
Flushing (Vascular disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (10) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 20 (28) | 7 (9)
Gastrointestinal disorders - Other, Abdominal cramping (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal disorders - Other, Bone sequestrum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Fractured tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, R upper jaw bone spicule (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Stomach virus (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Canker sore (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Cold Intolerance (General disorders) | 0 (0) | 2 (2)
General disorders and administration site conditions - Other, Foot cramps (General disorders) | 0 (0) | 1 (2)
General disorders and administration site conditions - Other, tooth fracture (General disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (15) | 8 (14)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 26 (116) | 19 (69)
Hemoglobinuria (Renal and urinary disorders) | 23 (91) | 22 (64)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 9 (11) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (9)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 13 (23) | 10 (22)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (54) | 13 (40)
Hyperkalemia (Metabolism and nutrition disorders) | 20 (57) | 12 (37)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (16) | 6 (10)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 7 (8) | 5 (5)
Hypertension (Vascular disorders) | 27 (49) | 15 (34)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperuricemia (Renal and urinary disorders) | 16 (63) | 5 (20)
Hypoalbuminemia (Metabolism and nutrition disorders) | 22 (102) | 23 (85)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (18) | 5 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 22 (65) | 12 (27)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (46) | 16 (38)
Hyponatremia (Metabolism and nutrition disorders) | 21 (97) | 19 (41)
Hypophosphatemia (Metabolism and nutrition disorders) | 22 (64) | 12 (27)
Hypotension (Vascular disorders) | 2 (2) | 5 (6)
Hypothyroidism (Endocrine disorders) | 11 (19) | 9 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infections and infestations - Other, Coronavirus (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Ear abscess (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Folliculitis R posterior thigh (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Infection R arm @ biopsy suture site (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Lyme Disease (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Pre auricular abscess (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, SARS COVID 2 POSITIVE (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Shingles (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Viral gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, Laceration to L 3rd phalange (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (14) | 11 (13)
Irregular menstruation (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Libido decreased (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Localized edema (General disorders) | 2 (2) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 17 (40) | 19 (52)
Lymphocyte count increased (Investigations) | 7 (21) | 3 (3)
Malaise (General disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Metabolism and nutrition disorders - Other, Night Sweats (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (13) | 4 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Achilles tendonitis L foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, BLE cramp (intermittent) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, BLE cramps at night (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Back spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Body aches/pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Groin strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, L foot heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, LLE leg/calf muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Leg cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Leg cramping/stiffness of feet (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle spasm, muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Muscle spasm-bilat lower abd (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Rib Pain-L posterior (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Thigh spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 4 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 (34) | 11 (15)
Nausea (Gastrointestinal disorders) | 22 (27) | 20 (25)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nervous system disorders - Other, Concussion (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Migraine headache (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Muscle twitches (intermittent) (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Tingling in bilateral hands/arms (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, nerve pain at surgical scar (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (10) | 2 (4)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 8 (9)
Oral dysesthesia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 4 (6) | 0 (0)
Pain (General disorders) | 13 (35) | 11 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (14) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 5 (5) | 2 (2)
Paronychia (Infections and infestations) | 20 (49) | 7 (12)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3)
Platelet count decreased (Investigations) | 10 (28) | 9 (24)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 38 (357) | 28 (149)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (15) | 9 (11)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 42 (80) | 35 (54)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Renal and urinary disorders - Other, Asymptomatic bacteria (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, Detrusor Sphincter Dyssynergia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 2 (3) | 3 (4)
Renal and urinary disorders - Other, Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal and urinary disorders - Other, Urinary hesitancy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, Hydrocele/scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, Labial sensitivity/soreness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, Vaginal spotting (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Serum amylase increased (Investigations) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 4 (6) | 7 (9)
Skin and subcutaneous tissue disorders - Other, Abrasion R ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Abscess R axilla (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Adhesive tape reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Angular Cheilitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Basal cell ca. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Bleeding gums (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Blepharitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Brittle nails (Skin and subcutaneous tissue disorders) | 14 (15) | 5 (6)
Skin and subcutaneous tissue disorders - Other, Chafing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cold sore (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Dry sinus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema eyelids (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Erythema flat rash L axilla/knee (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythematous painful groin rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Eczematous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Hair loss bilat hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Intermittent Mouth sores (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Intermittent tongue sores (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Inverse psoriasis of buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Lip sore; lower lip (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Lip ulcer/sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Melanotic macule buccal lesion R cheek (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Mouth blister/cold sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Mouth sore/swollen lip (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Mouth sores (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Mouth sores-intermittent (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Mouth sores/bleeding gums/stomatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Mucocutaneous disorder (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Nose Sores (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Pain around fingernails (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Periorbital erythema rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Poison Ivy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Psoriasiform hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other, R leg lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Reddened and irritated umbilicus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sensitivity & Tenderness under fingernails (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sores on bottom of feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Stye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sunburn (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Skin and subcutaneous tissue disorders - Other, Sunburn on face/upper torso (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Throat sores (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Tick bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Tinea cruris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Tinea corporis-breasts (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Tongue sores (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Skin and subcutaneous tissue disorders - Other, mouth sores (intermittent) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 12 (29) | 3 (6)
Skin ulceration (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Sore throat (Gastrointestinal disorders) | 9 (12) | 6 (6)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tooth discoloration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 10 (12) | 9 (14)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 2 (3) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (13) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 3 (3) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 16 (34) | 15 (27)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (20) | 10 (14)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 9 (26) | 3 (9)
Weight loss (Investigations) | 20 (78) | 14 (54)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 4 (8) | 4 (7)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT01130519/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT01130519/ICF_001.pdf